CLINICAL TRIAL: NCT06668779
Title: Digital Analysis of Tooth Crown Dimensions of Primary Teeth in a Group of Egyptian Children (4-6 Years) : (A Cross Sectional Study)
Brief Title: Digital Analysis of Primary Teeth Dimensions in a Group of Egyptian Children (4-6 Years)
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwan Magdy Abdelnaby Mohamed, dentist, Cairo University
Other Study IDs: Digital analysis of dimensions
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Digital Analysis of Tooth Crown Dimensions of Primary Teeth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Tooth size (Mesiodistal, Buccolingual and Occluso-gingival) has an important role in pediatric dentistry as it helps for fabrication of appropriate sizes of zirconia crowns for primary anterior teeth and Stainless-Steel crowns for primary posterior teeth. Tooth size differs among and within populations.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-6 years
2. Fully erupted first and second primary molars
3. Sound interproximal & buccal / lingual walls with or without minimal occlusal pits & fissure incipient caries.
4. No previous interproximal & buccal / lingual restorations
5. Intact mesial and distal marginal ridge

Exclusion Criteria:

1. Children with gross carious lesions.
2. Children with hypo-mineralization, hypoplasia and fracture.
3. Children with mental disability.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Egyptian children from the outpatient clinic of pediatric dentistry department Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
tooth crown dimensions of primary teeth | 8 months
  measurement of dimensions (Mesio-distal, Occluso-gingival and bucco-lingual) of primary anterior teeth and primary posterior teeth.

IPD SHARING:
Plan to Share IPD: Undecided